CLINICAL TRIAL: NCT03168906
Title: The RAIN Study, a Multicenter Randomized Double-blind Phase 2b Study of NEOD001 in Previously Treated Subjects With Systemic Light-chain (AL) Amyloidosis and Persistent Renal Involvement
Brief Title: Renal AL Amyloid Involvement and NEOD001
Acronym: RAIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOD001-RAIN
Record Dates: First submitted 2017-04-26; First posted 2017-05-30 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; NEOD001; RAIN
MeSH Terms: conditions — Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NEOD001 (Experimental): Study Drug given IV every 28 days at 24mg/kg
  Interventions: Drug: NEOD001
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NEOD001 — NEOD001 is a monoclonal antibody directed at soluble and insoluble light chain aggregates
  Arms: NEOD001
Drug: Placebo — Saline bag
  Arms: Placebo

SUMMARY:
This is a multicenter, Phase 2b, randomized, double-blind, placebo-controlled, two-arm, parallel-group efficacy and safety study of NEOD001 as a single agent administered intravenously in adults with AL amyloidosis who have a maintained hematologic response to their most recent treatment for AL amyloidosis (e.g., chemotherapy, autologous stem cell transplant [ASCT]) and have persistent renal dysfunction.

DETAILED DESCRIPTION:
This is a multicenter, Phase 2b, randomized, double-blind, placebo-controlled, two-arm, parallel-group efficacy and safety study of NEOD001 as a single agent administered intravenously in adults with AL amyloidosis who have a maintained hematologic response to their most recent treatment for AL amyloidosis (e.g., chemotherapy, autologous stem cell transplant [SCT]) and have persistent renal dysfunction. Subject screening will occur during the 28 days prior to the first administration of study drug (i.e. month 1 day 1). If screening assessments are completed and all eligibility requirements are met, the subject will be enrolled. Study visits will occur every 28 days based on scheduling from month 1 day 1. A ±5-day window is allowed for visits starting after month 1. Subjects may receive up to 12 infusions of study drug. Subjects who discontinue study drug before the initial End of Study (EOS) visit should have an Early Treatment Discontinuation (ETD) Visit 30 (±5) days after their final administration of study drug. After completing 12 months of treatment and the confirmatory EOS visit, a subject may enter an open-label extension (OLE) study, during which subjects will receive active treatment with NEOD001 for 12 months and may receive concurrent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Biopsy-proven diagnosis of AL amyloidosis by immunohistochemistry or mass spectroscopy of a tissue biopsy excluding bone marrow
3. Screening renal biopsy for RAIN confirming AL amyloidosis as exclusive or dominant cause of renal damage
4. Persistent renal involvement from diagnosis with proteinuria (predominantly albumin) > 500mg/day in a 24-hour urine collection
5. CKD 1 to 3 (eGFR > 30)
6. ≥1 prior systemic hematologic therapy for a free light chain (FLC) producing hematologic malignancy underlying the initial diagnosis of AL amyloidosis with at least a partial FLC response (PR, VGPR, CR) to treatment deemed stable and not requiring further treatment
7. ECOG Performance Status ≤ 2
8. Clinical laboratory values:

   1. Absolute neutrophil count > 1000/μL
   2. Platelet count > 75,000/μL
   3. Total bilirubin ≤ 1.5X ULN
   4. Alkaline phosphatase ≤ 5X ULN
   5. NT-proBNP < 1800 pg/mL
9. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care

Exclusion Criteria:

1. Amyloidosis due to mutations of the transthyretin gene or presence of other non-AL amyloidosis
2. Female patients who are lactating, breastfeeding, or pregnant
3. Patients who have not been treated or who have received chemotherapy within 6 months, or SCT within 12 months, for the light-chain producing hematologic disease causing AL amyloidosis, at the time of the first dose of NEOD001 (month 1 day 1)
4. Patients who at initial diagnosis or later met the International Myeloma Working Group (IMWG) definition of active multiple myeloma requiring therapy (Appendix 3)
5. Patients whose screening renal biopsies for RAIN show dominant causes of renal damage not related to AL amyloidosis
6. Medically documented cardiac syncope, uncompensated congestive heart failure, myocardial infarction within the previous 6 months, unstable angina pectoris, clinically significant repetitive atrial or ventricular arrhythmias despite antiarrhythmic treatment, or severe orthostatic hypotension or clinically significant uncompensated autonomic insufficiency
7. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
8. Ongoing or active infection, known HIV positive, known to be hepatitis B surface antigen-positive or has known or suspected active hepatitis C infection.
9. Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Comenzo, MD, Study Chair — Tufts Medical Center
Locations (9):
- United States (9):
  - Mayo Clinic- Arizona, Scottsdale, Arizona
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic- Florida, Jacksonville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic- Minnesota, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NEOD001 | Placebo
Started | 6 | 6
Completed | 0 (Study discontinued due to futile nature of drug) | 0 (Study discontinued due to futile nature of drug)
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEOD001 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 60 [47 to 78] | 54.5 [49 to 68] | 57.5 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Renal Response After Treatment With NEOD001
Description: A renal response is a ≥ 30% reduction in proteinuria in the absence of a ≥ 25% decrease in eGFR. A confirmed renal response is one that has been documented as present one month after 12 monthly treatments.
Time Frame: Baseline to 13 Months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Measured GFR at Study Entry
Description: The aim of this study is to assess the performance of CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) creatinine in comparison to iothalamate clearance measured in AL amyloidosis patients. Iothalamate will be given subcutaneously. Urine and plasma samples will then be obtained. All laboratory tests for samples obtained for GFR measurement will be performed at Mayo Clinic Rochester. Quantification of iothalamate in urine and plasma will be performed using a tandem mass spectrometric method.
Time Frame: Baseline
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to CKD 4 or 5
Description: Months to Chronic Kidney Disease level 4 or 5
Time Frame: Baseline to 13 Months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to eGFR ≤ 15 or Dialysis
Description: Months to estimated Glomerular Filtration Rate ≤ 15 or dialysis
Time Frame: Baseline to 13 Months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Doubling of Creatinine
Description: Months to doubling of serum creatinine
Time Frame: Baseline to 13 Months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to ≥ 40% Reduction in eGFR
Description: Months to ≥ 40% reduction in estimated glomerular filtration rate
Time Frame: Baseline to 13 Months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Renal Response in Patients With Maintained Hematologic Responses After 24 Monthly Treatments.
Description: A renal response is a ≥ 30% decrease in proteinuria or drop of proteinuria below 0.5 g/24h in the absence of renal progression.
Time Frame: Baseline to 26 months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: All Cause of Mortality at 26 Months
Description: Death at 26 months from Baseline due to any cause
Time Frame: Baseline to 26 months
Population: Trial was closed prior to completion, therefore data were not collected.
Arm/Group | NEOD001 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | NEOD001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NEOD001 (N=6) | Placebo (N=6)
Chest pain (General disorders) | 1 (1) | 0 (0)
Left arm pain (Nervous system disorders) | 1 (1) | 0 (0)
Right hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper and lower extremity swelling (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coughing spells (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03168906/Prot_SAP_000.pdf